CLINICAL TRIAL: NCT02210936
Title: Preventing Prescription Drug Problems: A Pilot Military Opioid Safety Initiative
Brief Title: SCOSI-M: Preventing Prescription Drug Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brandeis University (Other)
Collaborators: University of South Carolina (Other); Medical University of South Carolina (Other); Moncrief Army Community Hospital (Unknown); William Jennings Bryan Dorn VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14047
Record Dates: First submitted 2014-07-10; First posted 2014-08-07 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Prescription Drug Problems
MeSH Terms: interventions — Early Intervention, Educational

ARMS (1):
- PDMP Data (Other)
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — The design is primarily a pre-post, non-equivalent comparison group test of program effectiveness. If final sample size permits, we will examine program effects for each practice environment separately. For measures that require interview data there will be no comparison group data.
  We will construct matched comparison groups of physicians for each environment for which only secondary data analysis will be conducted. The matched comparison group will be constructed using prescription data from the DoD's pharmacy data transaction system (MACH and DORN VAMC) and from SCRIPTS (community-based physicians and VA prescribers).

SUMMARY:
Brandeis University and University of South Carolina (USC) have joined together to develop the South Carolina Opioid Safety Initiative - Military (SCOSI-M), to develop an academic detailing (medical education) intervention for physicians and evaluate its effectiveness in a pilot study. The goal of the intervention is to increase the use of safe prescribing and prescription monitoring practices among primary care physicians. The research team will design and pilot an educational intervention for physicians who treat military personnel, veterans, and their families with prescription opioids. The overall aim of SCOSI-M is to prevent the onset or progression of prescription drug problems among Iraq and Afghanistan veterans, military members, and their families who are at high risk for developing problems if their treatment involves long-term use of an opioid.

ELIGIBILITY:
Inclusion Criteria:

1. a physician within one of the 3 practice environments;
2. typically prescribes Schedule II opioids to 10 or more non-cancer pain patients each month;
3. if community office-based, a substantial number of patients must have TRICARE (e.g., 20%); and d) willing to provide written consent for data collection and release of own SCRIPTS data.

Exclusion Criteria:

1. non-physician providers who report data to the SCRIPTS (dentist, veterinarians, nurses),
2. surgeons, pediatricians, or physicians predominately treating pain in cancer or surgical patients, and,
3. not eligible to register as authorized SCRIPTS user.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-07; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Use of SCRIPTS | Up to 12 months
  Primary outcomes, or effectiveness, will be measured first by the use of SCRIPTS when prescribing opioids (e.g., % of new patients the physician queried; % of patients with long-term use the physician queried).

CONTACTS AND LOCATIONS:
Locations (1):
- Brandeis University, Waltham, Massachusetts, United States

REFERENCES:
- [Derived] Larson MJ, Browne C, Nikitin RV, Wooten NR, Ball S, Adams RS, Barth K. Physicians report adopting safer opioid prescribing behaviors after academic detailing intervention. Subst Abus. 2018;39(2):218-224. doi: 10.1080/08897077.2018.1449175. Epub 2018 May 4. PMID 29608412